CLINICAL TRIAL: NCT02203929
Title: Preoperative Progression of Macular Holes Using Optical Coherence Tomography
Brief Title: Preoperative Progression of Macular Holes
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Mark Alberti, BSc.med., Glostrup University Hospital, Copenhagen
Other Study IDs: MH-Progression
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Macular Holes
Keywords: Macular Holes; Progression
MeSH Terms: conditions — Retinal Perforations; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phakic eyes: Phakic eyes will be monitored with 4 preoperative optical coherence tomography scans as these patients will undergo phacoemulsification and intraocular lens implantation prior to their macular hole surgery
- Pseudophakic eyes: Phakic eyes will be monitored with 2 preoperative optical coherence tomography scans as there is no surgical intervention prior to the macular hole treatment.

SUMMARY:
Knowledge of the natural history and progression of macular holes is mainly limited to the studies from the pre-optical coherence tomography era. By observing macular holes preoperatively we are able to determine the extent of the preoperative macular hole progression.

At our institution macular holes are treated in an elective setting. The majority of macular holes undergo a 2-step sequence of phacoemulsification and intraocular lens implantation followed by vitrectomy.

We wish to observe the effect of time and cataract surgery on the progression of macular holes prior to vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic macular hole stage II-IV
* Informed consent
* Duration of symptoms ≤ 24 months

Exclusion Criteria:

* Previous vitreomacular surgery
* Ocular trauma
* Significant visual function affecting disease (proliferative diabetic retinopathy, diabetic macular edema, exudative macular degeneration)

Ages: 40 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Ophthalmic University Center
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Macular hole Progression | 3 months preoperative
  Serial optical coherence tomography (OCT) measurements in the preoperative period. The size of macular hole is determined by measuring the macular hole minimal linear diameter (µm).
  Size and stage of macular hole is determined at primary evaluation at tertiary ophthalmic center. Initial scan is followed by pre-vitrectomy scan if patient is pseudophakic. Initial OCT scan is followed by pre- and postcataract as well as pre-vitrectomy OCT scan if patient is pseudophakic.

SECONDARY OUTCOMES:
Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity | 3 months postoperative
  Visual acuity in ETDRS letters measured 3 month postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Morten la Cour, DMSc, Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Denmark